## Fascia of Scarpa in the formation of seroma in abdominoplasty after bariatric surgery.

Abdominoplasty after surgery to reduce stomach and weight loss, may develop a fluid in the abdominal wall (seroma) when leaving a layer of the abdominal wall called fascia.

It will be performed in 46 patients of the female genus anchor abdominoplasty. Divided into two groups of 23 patients. In one group the Scarpa fascia will be maintain and the other will not be maintained. All will use suction drain. The variables will be the total flow of the drain go while it remains, an amount of days of permanence. The drain will be withdrawn as the volume drained to less than 30 ml / 24 h. In the 20th postoperative day, abdominal wall ultrasound will be performed to diagnose seroma. Patients undergoing gastroplasty who need anchor abdominoplasty. Clinical trial of safety and efficacy, randomized, parallel, two-arm, blind.

## Inclusion criteria

Age between 25 and 55 years, Feminine gender, BMI less than 30 kg per m<sup>2</sup>, Not being nulliparous and at most three pregnancies, Without restriction as to ethnicity, schooling or social class, No smoking for at least 2 months.

## exclusion criteria

neoplasia, diabetes mellitus, systemic arterial hypertension diseases of the lymphatic system, and carriers of preexisting abdominal surgery scars, other than those resulting from bariatric surgery, and the Pfannenstiel scar.

The first 16 cases in each group were used as a pilot for the calculation of the sample. Fascia maintenance is expected to result in a 40% reduction in the amount of seroma and reduce at least 2 days in the use of the drain. With 80% power and 95% confidence, the required sample of women for the study should be 18 in each group, considering that the largest sample obtained was aimed at the difference in the amount of seroma. It was

observed that the mean volume in the group with preservation of the fascia was 249.1 ml, while the group without preservation presented a mean of 428.9, a statistically higher volume (p = 0.003) as evidenced by t-student test and Mann-whitney test.

verify if the measurements of the seroma differ according to the presence of scarpa fascia in 46 patients submitted to an abdominoplasty. All patients had the measurement of the drained liquid (seroma) in ml daily (volume of the drainage in 24 hours) by means of a closed suction drain.

A 20 ml syringe was used to measure the drained volume. Permanence on days with the drainage of the abdomen until the volume was less than 30 ml in 24 hours and volume of extracellular fluid in the subcutaneous (seroma) of abdominal wall measured by ultrasonography on the 20th postoperative day.

Permanence on days with the drainage of the abdomen until the volume was less than 30 ml in 24 hours and volume of extracellular fluid in the subcutaneous (seroma) of abdominal wall measured by ultrasonography on the 20th postoperative day

It was observed that the drainage time in patients with fascia preservation was on average 4.2 days, compared with 5.4 days in the fascia group, a significantly lower finding (p = 0.003). On the 20th postoperative day, the ultrasound volume was 16.8 ml in the preservation group and 21.6 ml without the fascia, statistically the same in the two groups of patients (p = 0.809), as evidenced by t-student test and mann-whitney test.